CLINICAL TRIAL: NCT01444651
Title: Phase 3 Randomized Trial of Tadalafil and Glycemic Traits
Brief Title: A Trial of Tadalafil and Glycemic Traits
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas J. Wang, MD (Other)
Responsible Party: Sponsor-Investigator, Thomas J. Wang, MD, Associate Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010P-001519
Record Dates: First submitted 2011-08-03; First posted 2011-10-03 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Cardiovascular Disease; Insulin Resistance; Glucose Intolerance; Obesity
Keywords: Tadalafil; Phosphodiesterase 5 Inhibitors; Cyclic Guanylyl Monophosphate Pathway; Pharmacologic Actions; Vasodilator Agents; Cardiovascular Agents; Obesity; Glycemic Traits; Insulin Resistance; Glucose Metabolism
MeSH Terms: conditions — Cardiovascular Diseases; Insulin Resistance; Glucose Intolerance; Obesity | interventions — Tadalafil; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Active Comparator): 20 mg Tadalafil tablet taken by mouth once a day for 3 months
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Placebo tablet taken by mouth once a day for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — 20 mg Tadalafil taken once a day for 3 months
  Other Names: Adcirca, Cialis
  Arms: Tadalafil
Drug: Placebo — Placebo tablet taken by mouth once a day for 3 months
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if tadalafil can help overweight and obese people metabolize blood sugar more efficiently. The investigators also want to find out if 20 mg/day of tadalafil for 3 months is safe to take without causing too many side effects. The investigators are plan to enroll 100 subjects at Massachusetts General Hospital (MGH).

DETAILED DESCRIPTION:
This study is examining changes in insulin resistance and glucose tolerance following 3 months of treatment with oral, once daily tadalafil.

The investigators primary hypotheses are that measurable decreases in insulin resistance (as measured by HOMA-IR) and increases in insulin sensitivity (as measured by the Matsuda index) will occur following 3 months of treatment with oral tadalafil 20 mg daily compared to placebo.

The investigators secondary hypotheses are that improvements in average glycemia (as measured by hemoglobin A1C), pancreatic beta cell function (as measured by the oral disposition index), and body composition (including weight, waist circumference, body mass index, and waist-hip ratio) will occur as a result of tadalafil-mediated changes in the cGMP pathway.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 50 years
* BMI > 30 kg/m2
* Fasting insulin > 10 uU/mL

Exclusion Criteria:

* Systolic blood pressure (SBP) < 100, > 150 mmHg
* Current anti-hypertensive medication use, including diuretics
* Current use of organic nitrates
* Current use of PDE-5 inhibitors (sildenafil, tadalafil, vardenafil)
* History of reaction to PDE-5 inhibitors
* Known HIV infection
* Use of medications that strongly alter CYP3A4 activity
* History of myocardial infarction, angina, uncontrolled cardiac arrhythmia, stroke, transient ischemic attack, or seizure
* Known non-arteritic ischemic optic retinopathy (NAIOR)
* History of hearing loss
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2 by the modified diet in renal disease (MDRD) equation
* Hepatic transaminase (AST and ALT) levels greater than three times the upper limit of normal
* Known pregnancy or those unwilling to avoid pregnancy during the course of the study
* History of priapism
* Use in excess of four alcoholic drinks daily
* History of diabetes mellitus or use of anti-diabetic medications
* Known anemia (men, Hct < 38% and women, Hct < 36%)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Wang, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ho JE, Arora P, Walford GA, Ghorbani A, Guanaga DP, Dhakal BP, Nathan DI, Buys ES, Florez JC, Newton-Cheh C, Lewis GD, Wang TJ. Effect of phosphodiesterase inhibition on insulin resistance in obese individuals. J Am Heart Assoc. 2014 Sep 11;3(5):e001001. doi: 10.1161/JAHA.114.001001. PMID 25213566

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 111 participants screened, 38 excluded (34 did not meet eligibility criteria, 2 unable to obtain intravenous access, 2 withdrew consent)
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 36 | 37
Completed | 25 | 28
Not Completed | 11 | 9
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 5 | 5
Not completed — Non-fasting | 2 | 1
Not completed — Missing data | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9) | 34 (9) | 33 (9)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 18 | 15 | 33
Region of Enrollment [Number; unit: participants]
  United States | 25 | 28 | 53
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 38.7 (6.8) | 36.8 (6.8) | 37.7 (6.8)
Fasting insulin [Mean (Standard Deviation); unit: microunits/mL] | 17 (10) | 17 (16) | 17 (13)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Resistance From Baseline to 3 Months, as Measured by HOMA-IR
Description: The primary endpoint is defined as the treatment group difference in the change in insulin resistance (baseline HOMA-IR minus 3-month HOMA-IR). HOMA-IR = [fasting glucose * fasting insulin]/405
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg*microunits/dL*mL
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 25 | 28
mg*microunits/dL*mL
  Baseline | 3.57 (2.86) | 3.84 (3.80)
  3 months | 3.81 (5.14) | 5.06 (3.95)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Linear regression was used to model the change in HOMA-IR (3 month minus baseline value), comparing tadalafil versus placebo groups after adjusting for baseline HOMA-IR; Test type: Superiority or Other; p = 0.34, Regression, Linear; beta estimate = -1.25, Standard Error of Mean 1.29

2. Secondary Outcome: Baseline to 3-month Change in Insulin Sensitivity, as Measured by the Matsuda Index
Description: The secondary endpoint is defined as the treatment group difference in the change in Matsuda Index (baseline minus 3-month). This index is a measure of insulin resistance derived from a frequently sampled oral glucose tolerance test, obtaining glucose and insulin levels in the fasting state, as well as 30, 60, 90, and 120 min after administration of oral glucose load. Matsuda index = 10,000/SQRT [fasting glucose*fasting insulin* (mean glucose from time 30, 60, 90, 120 min) * (mean insulin at time 30, 60, 90, and 120 min)]
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: unitless index
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 25 | 28
unitless index
  Baseline | 3.60 (2.54) | 3.51 (2.15)
  3 months | 4.27 (2.83) | 3.28 (2.42)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Linear regression was used to model the change in Matsuda Index (3-month minus baseline), comparing tadalafil versus placebo groups after adjusting for baseline value; Test type: Superiority or Other; p = 0.18, Regression, Linear; beta estimate = 0.96, Standard Error of Mean 0.68

3. Secondary Outcome: Baseline to 3-month Change in Endothelial Function Measured by EndoPAT
Description: Endothelial function was measured using the reactive hyperemia index, acquired using EndoPAT device. Peripheral arterial tonometry probes were placed on both index fingers. After a 5 min equilibration period, a blood pressure cuff was inflated to 200 mmHg and kept inflated for 5 min. The cuff was then rapidly deflated and the reactive hyperemic response pulse volume recorded, where RHI = ratio of hyperemic finger pulse volume (post-cuff inflation / pre-cuff inflation) to control finger pulse volume (post-cuff inflation / pre-cuff inflation)
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: unitless index
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 25 | 28
unitless index
  Baseline | 2.1 (0.5) | 2.3 (0.6)
  3-month | 2.1 (2.7) | 2.2 (0.3)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Linear regression was used to model the difference in EndoPAT (3-month minus baseline), comparing tadalafil to placebo groups after adjusting for baseline values; Test type: Superiority or Other; p = 0.76, Regression, Linear; beta estimate = -0.18, Standard Error of Mean 0.58

4. Secondary Outcome: Insulinogenic Index
Description: The secondary endpoint is defined as the treatment group difference in the change in insulinogenic index (baseline minus 3-month). This index is thought to reflect insulin secretion, and is derived from fasting and 30 min-post oral glucose tolerance testing glucose and insulin values. Insulinogenic index = [fasting insulin - insulin at time 30 min] / [fasting glucose - glucose at time 30 min]
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: unitless index
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 25 | 28
unitless index
  Baseline | 0.39 (8.04) | 2.17 (2.06)
  3-month | 2.62 (3.03) | 1.04 (2.32)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Linear regression was used to model the change in insulinogenic index (3-month minus baseline), comparing tadalafil to placebo groups after adjusting for baseline value; Test type: Superiority or Other; p = 0.06, Regression, Linear; beta estimate = 1.48, Standard Error of Mean 0.77

5. Secondary Outcome: Baseline to 3 Month Change in Composite of Insulin Resistance and Sensitivity, as Measured by the Oral Disposition Index
Description: The secondary endpoint is defined as the treatment group difference in the change in oral disposition index (baseline minus 3-month). This is thought to reflect a composite of both insulin resistance and secretion. Oral disposition index = insulinogenic index / fasting insulin
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: unitless index
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 25 | 28
unitless index
  Baseline | 1.74 (11.56) | 2.87 (3.67)
  3-month | 4.48 (4.62) | 0.58 (5.21)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Linear regression was used to model the change in oral disposition index (3-month minus baseline), comparing tadalafil versus placebo groups after adjusting for baseline value; Test type: Superiority or Other; p = 0.009, Regression, Linear; beta estimate = 3.76, Standard Error of Mean 1.38

6. Secondary Outcome: Baseline to 3-month Change in Matsuda Disposition Index
Description: Change in disposition index from baseline to 3 months. This index is a composite measure thought to reflect insulin resistance and secretion. Matsuda disposition index = [Matsuda sensitivity index * insulinogenic index]
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: unitless index
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 25 | 28
unitless index
  Baseline | 2.23 (24.19) | 6.67 (9.45)
  3-month | 9.22 (8.51) | 0.19 (18.42)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Linear regression was used to model the change in Matsuda disposition index (3-month minus baseline), comparing tadalafil to placebo groups after adjusting for baseline value; Test type: Superiority or Other; p = 0.05, Regression, Linear; beta estimate = 8.09, Standard Error of Mean 4.05

ADVERSE EVENTS:
Time Frame: Adverse events recorded during study duration (3 months)
Description: Adverse events ascertained at each follow-up visit
Arm/Group | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 7/36 | 2/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tadalafil (N=36) | Placebo (N=37)
Headache (Vascular disorders) | 4 | 0
Blurry vision and headache (Vascular disorders) | 0 | 1
Back or leg pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache and back ache (Musculoskeletal and connective tissue disorders) | 1 | 0
arm pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No